CLINICAL TRIAL: NCT00088387
Title: Glycogen Synthetase Kinase 3 (GSK-3) Inhibition in Alzheimer's Disease
Brief Title: Effect of Lithium and Divalproex in Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040243; 04-N-0243
Record Dates: First submitted 2004-07-23; First posted 2004-07-26 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-03

CONDITIONS: Alzheimer Disease
Keywords: Tau; T181; T231; Amyloid Beta; Beta-Catenin; Alzheimer Disease; AD
MeSH Terms: conditions — Alzheimer Disease; Pick Disease of the Brain; Plaque, Amyloid | interventions — Valproic Acid; Lithium

INTERVENTIONS:
Drug: Divalproex
Drug: Lithium

SUMMARY:
This study will examine the effect of the drugs lithium and divalproex (Depakote) on tau proteins, a type of protein in the brain and spinal fluid that are altered in patients with Alzheimer's disease. Both drugs are approved by the Food and Drug Administration to treat mood disorders, and both have been shown in animal studies to decrease the amount of altered tau protein. This study will determine whether lithium alone or in combination with divalproex reduces the altered tau protein in the spinal fluid of patients with Alzheimer's disease.

Patients with Alzheimer's disease who are between 40 and 90 years of age may be eligible for this study. Candidates are screened with a medical history and physical examination, neurologic and neuropsychological evaluation, blood and urine tests, electrocardiogram (EKG), and, if needed, a magnetic resonance imaging (MRI) scan of the brain.

Participants undergo the following tests and procedures:

* Drug treatment: Patients take study drugs for 6 weeks.
* Weekly clinic visits: Patients come to the clinic once a week for a physical examination, blood and urine tests, a review of drug side effects, and to receive the next week's supply of medications.
* Lumbar puncture (spinal tap): Patients have a lumbar puncture at study weeks 2, 4, and 6 to measure various brain chemicals and tau proteins in the cerebrospinal fluid (CSF), which bathes the brain and spinal cord. For this test, a local anesthetic is given and a needle is inserted in the space between the bones in the lower back where the CSF circulates below the spinal cord. A small amount of fluid is collected through the needle.
* Follow-up visit: Two weeks after completing the study medication, patients return to the clinic for a final evaluation, including a physical examination and blood and urine tests.

DETAILED DESCRIPTION:
The overall objective of this study is to examine the acute effects of lithium alone and/or in combination with divalproex on surrogate measures of neuroprotective activity in patients with Alzheimer's disease. It is hypothesized that at safe and tolerable doses these drugs will inhibit glycogen synthase kinase-3 activity and reduce the phosphorylated tau epitopes threonine-181 and threonine-231 implicated in the pathogenesis of this disorder. In this proof-of-principle study, efficacy on reducing tau phosphorylated epitopes will be assessed through cerebrospinal fluid (CSF) measurements. Safety will be monitored by means of frequent clinical evaluations and laboratory tests.

ELIGIBILITY:
INCLUSION CRITERIA:

Patient is between the ages of 40 and 90 (inclusive).

Patient will have a diagnosis of AD; the study will be confined to patients who are able to provide consent (pass a capacity assessment).

The modified Hachinski Ischemia Score must be less than 4.

Brain MRI performed within 15 months of enrollment must be compatible with the diagnosis of AD.

Patient and/or caregiver are willing to adhere to protocol requirements as evidenced by written, informed consent.

EXCLUSION CRITERIA:

Patients meeting any of the following exclusion criteria during screening or during the study will not be enrolled or will be immediately excluded from the study, as appropriate:

Patient has a history of any medical condition that can reasonably be expected to subject the patient to unwarranted risk.

Patient has clinically significant laboratory abnormalities that would preclude administration of lithium and divalproex.

Patient is taking a prohibited concomitant medication. The following medications are forbidden for at least one month prior to the treatment phase (unless otherwise noted) and during the course of the study:

Any investigational drugs;

Anti-depressants (eligibility will be considered as long as dosage remains stable throughout the study);

Anticonvulsants and other mood stabilizing drugs;

Treatment that may provoke lithium toxicity due to reduced renal clearance, including metronidazole, spectinomycin, tetracycline;

Treatment that may substantially increase steady-state plasma lithium levels resulting in lithium toxicity, including angiotensin-converting enzyme inhibitors, NSAIDS, diuretics;

Treatment that may increase the risk of neurotoxicity, including calcium channel blocking agents;

Drugs that may increase urinary lithium excretion resulting in lower serum lithium concentrations, such as acetazolamide, urea, xanthine preparations, alkalinizing agents such as sodium bicarbonate, theophylline;

Drugs that interact with lithium, including methyldopa;

Neuroleptics (eligibility will be considered as long as dosage remains stable throughout the study). If patient is on existing atypical neuroleptic drugs, these will be continued at the same dose. Patients will not start a new prescription for atypical antipsychotics during the study;

Drugs that may prolong the effects of lithium, including neuromuscular blocking agents;

Digoxin, warfarin.

Patient has not been using an adequate contraceptive method for the last 30 days or unwilling to continue contraception throughout the study, or is not at least one year post-menopausal (if female).

Patient is pregnant or breastfeeding.

Patient has participated in a clinical study with an investigational drug within the last 30 days.

Patient has a condition (such as active drug or alcohol abuse) that, in the opinion of the investigators, would interfere with compliance or safety.

Patient has known hypersensitivity to lithium or divalproex.

Patient's inability to swallow tablets or to comply with medication schedule.

Patient has no adequate caregiver.

Patient and/or caregiver are unwilling to sign an informed consent or to comply with protocol requirements.

Patient is unwilling to have lumbar puncture.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35
Dates: Start 2004-07; Study Completion 2005-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Bloom BS, de Pouvourville N, Straus WL. Cost of illness of Alzheimer's disease: how useful are current estimates? Gerontologist. 2003 Apr;43(2):158-64. doi: 10.1093/geront/43.2.158. PMID 12677073
- [Background] Knopman D. Pharmacotherapy for Alzheimer's disease: 2002. Clin Neuropharmacol. 2003 Mar-Apr;26(2):93-101. doi: 10.1097/00002826-200303000-00009. PMID 12671529
- [Background] Arai H, Terajima M, Miura M, Higuchi S, Muramatsu T, Machida N, Seiki H, Takase S, Clark CM, Lee VM, et al. Tau in cerebrospinal fluid: a potential diagnostic marker in Alzheimer's disease. Ann Neurol. 1995 Oct;38(4):649-52. doi: 10.1002/ana.410380414. PMID 7574462